CLINICAL TRIAL: NCT04194359
Title: Evaluation on the Tolerance and Preliminary Efficacy of Sintilimab (IBI308) Combined With Bevacizumab, Oxaliplatin and Capecitabine Regimen for Ras Gene Mutant and Microsatellite Stable Unresectable Metastatic Colorectal Cancer
Brief Title: Sintilimab (IBI308) Combined With Bevacizumab + XELOX Regimen in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-552
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Colorectal Cancer; RAS Mutation; Microsatellite Stable
Keywords: RAS-mutant Metastatic Colorectal Cancer; Immunotherapy; Anti-PD-1; Checkpoint; Efficacy; Safety; Microsatellite stable
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab (IBI308) plus Bevacizumab, Oxaliplatin and Capecitabine (Experimental): Sintilimab (IBI308)：200MG, once every three weeks; Bevacizumab:7.5mg/kg, once every three weeks; oxplatin: 135 mg per square meter body surface, once every three weeks; Capecitabine : Capecitabine 1 gram per square meter body surface area, from the first day to the 14th day
  Interventions: Drug: Sintilimab (IBI308)+bevacizumab+oxaliplatin+capecitabine

INTERVENTIONS:
Drug: Sintilimab (IBI308)+bevacizumab+oxaliplatin+capecitabine — Humanized PD-1 antibody (Sintilimab, IBI308)+bevacizumab+oxaliplatin+capecitabine

SUMMARY:
A phase II clinical study of Sintilimab (IBI308) combined with Bevacizumab, Oxaliplatin and Capecitabine regimen as first-line treatment in patients with RAS-mutant and microsatellite stable metastatic colorectal cancer. A total of 25 patients are planned to be enrolled.

DETAILED DESCRIPTION:
This study is a phase II clinical study of Sintilimab (IBI308) combined with bevacizumab + XELOX regimen as first-line treatment in patients with RAS-mutant and microsatellite stable metastatic colorectal cancer. The study treatment took 21 days as a treatment cycle. Sintilimab (IBI308), bevacizumab and oxaliplatin were given intravenously on the first day of each cycle, and capecitabine was given from the first day to the 14th day. All adverse events will be graded according to NCI CTCAE (version 5.0). Up to 8 courses of inductive therapy would be given. During the treatment, CT was rechecked every 2 courses to evaluate the curative effect. Patients with objective response or stable disease (SD) would continue to receive sintilimab plus bevacizumab and oral capecitabine in each 21-day cycle as maintenance therapy until the confirmation of disease progression, death, unacceptable toxicity, or withdrawal of consent.

A total of 25 patients are planned to be enrolled. When the number of subjects reaches 25 respectively, the enrollment ends to inquire about the safety and efficacy of Sintilimab (IBI308) combined with bevacizumab + XELOX.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years old, ≤ 75 years old;
2. Metastatic colorectal adenocarcinoma confirmed by histology and unresectable metastatic colorectal cancer confirmed by a multidisciplinary team;
3. RAS gene mutation, BRAF wild-type and microsatellite stable confirmed by polymerase chain reaction using a panel of six mononucleotide repeat markers (BAT-25, BAT-26, NR-21, NR-24, NR-27, and MONO-27);
4. ECOG performance status of 0-1;
5. Life expectancy≥3 months;
6. Adequate organ and bone marrow functions: absolute neutrophil count >1.5×109/L, hemoglobin >8 g/dL, platelet count >100×109/L, prothrombin time <1.5 upper limit of normal (ULN), activated partial thromboplastin time <1.5 ULN, bilirubin ≤1.5×ULN (could be extended to 3×ULN in case of liver metastasis), blood aspartate aminotransferase and alanine aminotransferase ≤2.5×ULN (could be extended to 5×ULN in case of liver metastasis), serum creatinine level ≤1.5×ULN or creatinine clearance ≥50 mL/min, urinary protein / creatinine ratio < 1 (or urine analysis < 1 + or 24-hour urinary protein < 1g / 24 h;
7. Informed consent has been signed;
8. The presence of at least one measurable lesion assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;

Exclusion Criteria:

1. received previous treatment with any anti-programmed cell death protein 1 (PD-1) or anti-PD-L1 antibody;
2. received treatment with corticosteroids or other immunosuppressive agents within 14 days prior to study drug administration;
3. presence of autoimmune disease, known interstitial lung disease;
4. those with previous or concurrent malignancies expect for basal cell carcinoma, cutaneous squamous cell carcinoma, or cervical carcinoma in situ that have undergone radical treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From Baseline to disease progress, up to 18 months
  Objective Response Rate was defined as the proportion of patients with a best objective response of complete response (CR) or partial response (PR) according to RECIST criteria (version 1.1).
Adverse Events and Serious Adverse Events | From Baseline to primary completion date, about 2 years
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.

SECONDARY OUTCOMES:
Disease Control Rate | From Baseline to disease progress, up to 18 months
  Disease Control Rate was defined as the proportion of patients with CR, PR, or SD according to RECIST criteria (version 1.1)
Progression free survival | From Baseline to primary completion date, about 2 years
  Progression-free survival is defined as the time from enrollment to the first documented disease progression according to RECIST version 1.1, or to death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, MD, Study Chair — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Fang X, Zhu N, Zhong C, Wang L, Li J, Weng S, Hu H, Dong C, Li D, Song Y, Xu D, Wang J, Sun L, Wang J, Wang Z, Cao H, Liao X, Yu N, Xiao Q, Mi M, Zhang S, Ding K, Yuan Y. Sintilimab plus bevacizumab, oxaliplatin and capecitabine as first-line therapy in RAS-mutant, microsatellite stable, unresectable metastatic colorectal cancer: an open-label, single-arm, phase II trial. EClinicalMedicine. 2023 Jul 27;62:102123. doi: 10.1016/j.eclinm.2023.102123. eCollection 2023 Aug. PMID 37554125